CLINICAL TRIAL: NCT02039284
Title: Efficacy of New Protocols in the Treatment of Upper Limb Dysfunctions in Patients With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101-5261A3
Record Dates: First submitted 2013-09-18; First posted 2014-01-17 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2017-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; novel intervention; sensory electrical stimulation; virtual reality; cycling training; constraint-induced therapy; biomechanical; physiology; outcome
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SES group (Experimental): SES group received the SES training in addition to traditional rehabilitation. Each SES session involved electrical stimulation followed by UE training in addition to home program.
  Interventions: Device: SES
- VCT group (Experimental): VCT group received the VCT training in addition to traditional rehabilitation.Each UE VCT session involved upper limb cycling training followed by UE training in addition to home program. The cycling program consisted of a warm-up exercise, twenty repetitions of hand push-up movements in the sitting position, UE cycling, and a cool-down exercise.
  Interventions: Device: VCT
- VRCIT group (Experimental): VRCIT group received the VRCIT training in addition to traditional rehabilitation.Each VRCIT session involved practice of functional tasks with the more affected UE followed by virtual-reality based eye-hand coordination tasks with the more affected UE for, in addition to home program, and restraint of the less affected UE for 3.5 to 4 hours per day.
  Interventions: Device: VRCIT
- traditional rehabilitation group (Active Comparator): Shame control group received the shame SES and traditional rehabilitation programs.
  Interventions: Device: traditional rehabilitation program

INTERVENTIONS:
Device: SES — SES group received the SES training in addition to traditional rehabilitation. Each SES session involved electrical stimulation followed by UE training in addition to home program.The novel SES programs were conducted three times per week, for 12 weeks. Each SES session involved electrical stimulation followed by UE training in addition to home program. The SES was applied to the forearm and whole hand with mesh glove for 20-30 minutes and arm with wrap for 20-30 minutes. The pulse width was set to 300 us for all stimulation levels. The frequency was set to 40-50 Hz.
  Other Names: novel sensory electrical stimulation program
  Arms: SES group
Device: VCT — The UE VCT programs were conducted three times per week, for 12 weeks. Each UE VCT session involved upper limb cycling training followed by UE training in addition to home program. The cycling program consisted of a warm-up exercise, twenty repetitions of hand push-up movements in the sitting position, UE cycling, and a cool-down exercise. The warm-up and cool-down exercises involved stretching and relaxing the head, neck, and the upper and lower body.
  Other Names: The upper extremity programsvirtual cycling training program
  Arms: VCT group
Device: VRCIT — VRCIT group received the VRCIT training in addition to traditional rehabilitation, conducted three times per week, for 12 weeks. Each VRCIT session involved practice of functional tasks with the more affected UE followed by virtual-reality based eye-hand coordination tasks with the more affected UE for, in addition to home program, and restraint of the less affected UE for 3.5 to 4 hours per day. The functional training of the more affected UE focused on massive practice of functional activities using the more affected arm, with the principles of shaping and repetitive task practice applied during training.
  Other Names: virtual reality based Constraint-induced therapy
  Arms: VRCIT group
Device: traditional rehabilitation program — The absence of muscle contractions was controlled by the investigator the sham stimulation was carried out identically, but the stimulation amplitude was set to 0 milliampere(mA). Subjects were not informed about the stimulation level and were instructed to distract attention from the stimulation.
  Arms: traditional rehabilitation group

SUMMARY:
Cerebral palsy (CP) is the most common childhood motor disability. Weakness, spasticity, and loss of dexterity are the major problems in patients with CP. A novel virtual cycling training (VCT) program for lower limb was to enhance promising muscle strength through promoting the participant compliance and motivation. Sensory electrical stimulation(SES) of whole hand is a novel technique and is commonly used to treatment of spasticity for patients with stroke. Constraint-induced therapy (CIT) is a method for treating developmental disregard and learned non-use of affected limb and improving motor efficiency, functional performance, and activities of daily living for patients with CP.

DETAILED DESCRIPTION:
This study will proposed 3 novel protocols, including upper extremity (UE) VCT, UE SES, and virtual reality based CIT (VRCIT) in the treatment of upper limb dysfunction in patients with CP. investigators hypothesize that the functioning and health-related quality of life (HRQOL) will improve through biomechanical and physiological changes after different treatment protocols in patients with CP. The biomechanical and physiological changes varied depending on different treatment protocols. This project aims to: 1. the immediate effects of new protocols in these patients through biomechanical, physiological, and clinical measures; 2. the maintaining effects of new protocols in these patients through biomechanical, physiological, and clinical measures;3. the most effective treatment protocol; 3. the biomechanical and physiological mechanism underlying clinical improvement; and 5. the clinical predictors influencing the outcome for new protocols.

This 4-year project will recruit an estimated 92-100 patients with CP. A blind, randomized controlled trial (RCT) study was designed. In the phase I (1st year), investigators will set-up the experimental protocols and perform pilot study. Twenty patients will be randomized into 4 groups: SES, VCT, VRCIT, and shame control groups. In the phase II (2nd -3rd year), 36-40 patients will be randomized into 2 groups: SES and shame control groups. In the phase III (3rd -4th year), 36-40 patients will be randomized into 2 groups:VCT and VRCIT groups. The outcome measures include biomechanical, physiological (muscle tone, muscle strength and endurance, kinematics, bone density, body compositions, metabolism), and clinical assessments, including functioning (motor impairment, movement and participation) and HRQOL, based on the International Classification of Functioning, Disability and Health (ICF) framework. The outcome measures will be administered at before, immediately after 12-week intervention, and 3-month follow-up assessments.

This project is significant for the translational and evidence-based medicine on CP neurorehabilitation. The research will offer valuable biomechanical and physiological biomarker that support motor control models proposed to account for motor problems and new protocol intervention in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis with spastic CP with Gross Motor Function Classification System(GMFCS) levels I-IV
2. aged 3-20 years
3. ability to undergo clinical assessment
4. ability to comprehend commands and cooperate during an examination

Exclusion Criteria:

1. chromosomal abnormalities
2. progressive neurological disorder or severe concurrent illness or disease not typically associated with CP
3. active medical conditions such as pneumonia or poor physical conditions that would interfere with participation
4. any major surgery or nerve block in the preceding 3 months
5. metabolic or hormonal disturbance
6. cardiovascular disorder
7. poor tolerance or a poor cooperation during assessment

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
change from baseline of muscle tone of the upper limb muscles in 12 and 24 weeks | baseline, 12weeks, 24weeks
  muscle tone of the upper limb muscles assessment by Modified Ashworth Scale and Myoton( © 2011 Myoton AS.).
change from baseline of Basic motor abilities in 12 and 24 weeks | baseline, 12 weeks, 24 weeks
  Basic motor abilities included the assessments of the Bruininks- Oseretsky Test of Motor Proficiency II (BOT II), Melbourne Assessment 2 (MA2), Quality of upper extremity skills test (QUEST). The measure is a composite.

SECONDARY OUTCOMES:
change from baseline of basic motor functions in 12 and 24 weeks | baseline, 12weeks, 24weeks
  Basic motor functions included the assessments of the Beery-Buktenica Developmental Test of Visual-Motor Integration (VMI-Chinese), Test of Visual Perceptual Skills, third edition, (TVPS-3), Sensory profile (SP)-Chinese.The measure is a composite.
change from baseline of quality of life in 12 and 24 weeks | baseline, 12weeks, 24weeks
  The health-related quality of life(HRQOL) assess by Cerebral Palsy Quality of Life (CP QOL) for Child and adolescent. The CP QOL is a measure of HRQOL specific to children and adolescent with cerebral palsy.
change from baseline of activities of daily living (ADL) in 12 and 24 weeks | baseline, 12weeks, 24weeks
  The ADL assessments included Functional Independence Measure for Children (WeeFIM), Pediatric Motor Activity Log (PMAL), etc.. The measure is a composite.
change from baseline of participation in 12 and 24 weeks | baseline, 12weeks, 24 weeks
  The assessments for participation included Assess of Preschool Children's Participation(APCP), Children Assessment of Participation and Enjoyment(CAPE) and Preferences for Activity of Children(PAC), and Adaptive Behavior Assessment System, second edition(ABAS-II)-Chinese, etc..The measure is a composite.
change from baseline of bone mineral density in 12 and 24 weeks | baseline, 12weeks, 24weeks
  The areal bone mineral density (aBMD) (g/cm2) will be measured at the lumbar spine (L1 to L4) and the humerus of the more-affected limb using dual X-ray absorptiometry (DXA).
change from baseline of Metabolism and Body composition in 12 and 24 weeks | baseline, 12weeks, 24weeks
  The measure included the total energy expenditure (kcal/min), active energy expenditure (kcal/min), total number of steps, physical activity levels and duration, sleep duration and efficiency, weight, total body water, skeletal muscle mass (SMM), body fat mass (BFM), fat free mass, percent body fat, waist-hip ratio (WHR), and basal metabolic rate (BMR) by the devices of SenseWear(© 2013 BodyMedia, Inc.) and Body Composition Analyzer(InBody220). The measure is a composite.
change from baseline of kinematic analysis in 12 and 24 weeks | baseline, 12weeks, 24weeks
  Kinematic analysis for patients performing Reach-to-grasp and Eye-hand coordination tasks.The measure is a composite.
change from baseline of muscle strength and endurance in 12 and 24 weeks | baseline, 12 weeks, 24 weeks
  Measure muscle strength and endurance by the device which combines range of motion, muscle testing (MicroFET3) and grip and pinch gauge (MicroFET 4) and data capture software.
change from baseline of severity in 12 and 24 weeks | baseline, 12 weeks, 24 weeks
  The severity is evaluated by Gross Motor Function Classification System(GMFCS), Manual Ability Classification System (MACS).The assessments for body function included Modified Ashworth Scale (MAS), strength, endurance, and trunk and limb involvement, etc. The measure is a composite.
change from baseline of reaction-time in 12 and 24 weeks | baseline, 12 weeks ,24 weeks
  To examine the reaction time by CANTAB® software.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD,PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No